CLINICAL TRIAL: NCT02499094
Title: Modeling and Predicting Real World Behavior Using Mobile Sensor Data on Patients With Major Depressive Disorder: Protocol for a Randomized Controlled Study
Brief Title: Modeling and Predicting Real World Behavior Using Mobile Sensor Data on Patients With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ginger.io (Industry)
Responsible Party: Principal Investigator, Gourab De, Data Scientist, Ginger.io
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GIO-001
Record Dates: First submitted 2015-07-14; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention A- Heuristic based (Experimental): Behavioral-data driven support, both mobile phone application and phone-based, informed by their self-reported symptom assessment as well as simple heuristic-based behavioral measures
  Interventions: Other: Behavioral-data driven support
- Intervention B- Machine Learning Based (Experimental): Behavioral-data driven support, both mobile phone application and phone-based, informed by their self-reported symptom assessment as well as machine learning model-based behavioral measures
  Interventions: Other: Behavioral-data driven support
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Behavioral-data driven support — Phone-based support (e.g. triaging of the situation, emotional support, and guidance on next steps for the patient) and in-app support (health education content based on cognitive behavioral therapies, mindfulness, and behavioral activation)
  Arms: Intervention A- Heuristic based; Intervention B- Machine Learning Based

SUMMARY:
The purpose of this study is to validate the effectiveness of using an integrated mobile sensing platform to deliver large-scale data-driven interventions to patients with depression.

DETAILED DESCRIPTION:
This study is a smartphone-based, randomized, single-blind, controlled parallel-

design study with two intervention arms and one control arm. The two intervention arms

will receive in-app messages and phone-based support, which will be triggered by

participant's self-reported surveys and passive behavioral data gathered through a

smartphone app. The study will include a nationwide sample of adult (18 years or older)

smartphone users, who are currently experiencing depressive symptoms. The primary

outcome will be decrease in depression symptom severity, as measured by the 9-item

Patient Health Questionnaire, over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Currently suffering from depression (as measured by a PHQ-9 score of 10 or more at the time of screening)
* Own an iPhone or Android smartphone with a mobile voice calling plan with a US carrier
* Fluency in English

Exclusion Criteria:

* Participants with visual or hearing impairment
* Recent history of pregnancy (currently pregnant or those who have given birth within the past four months at the time of screening)
* Recent loss of a loved one (within the past two months at the time of screening)
* Unable or unwilling to accept End User License Agreement, or to provide information regarding their demographic characteristics and mental health history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1004 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in depression symptom severity | 6 months
  Change in the 9-item Patient Health Questionnaire (PHQ-9) score from baseline

SECONDARY OUTCOMES:
Change in patient activation | 6 months
  Change in the 13-item Patient Activation Measure score from baseline